CLINICAL TRIAL: NCT00748293
Title: Achievement of Better Examinee Compliance on Colon Cleansing Before Colonoscopy Without Sacrificing Cleansing Effect - A Multi-Center Endoscopist-Blinded Randomized Trial Using Commercialized Low-Residue Diet
Brief Title: Achievement of Better Examinee Compliance on Colon Cleansing Using Commercialized Low-Residue Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Medical University Hospital (Other); E-DA Hospital (Other); Buddhist Tzu Chi General Hospital (Other); En Chu Kong Hospital (Other)
Responsible Party: Han-Mo Chiu, National Taiwan Univesity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 200802030R
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2008-09

CONDITIONS: Colonoscopy; Colon Cleansing; Low-Reside Diet
Keywords: Colonoscopy; Colon cleansing; Low-reside diet; Compliance; PEG-ELS
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention): PEG-ELS 2000 ml ingestion in the morning of colonoscopy
- B (Other): Low-reside diet on previous day (breakfast, lunch and dinner), PEG-ELS 1500 mL in the morning of colonoscopy
  Interventions: Other: Low-residue diet

INTERVENTIONS:
Other: Low-residue diet — Commercialized (not yet marketed)low-residue diet
  Arms: B

SUMMARY:
Good colon cleansing is pivotal for achieving speedy and safe colonoscopic examination with high adenoma detection rate.Previous studies, including our previous RCT conducted in 2004 to 2005, have demonstrated that high yield rate can be achieved by on-the-day colon preparation with 2000 ml PEG-ELS. Poor patient compliance, however, is the main hurdle to complete ingestion of 2000 ml PEG-ELS not only for subjects with lower body weight but also for those with normal BMI or body weight.The main cause of poor patient compliance includes abdominal pain, bloating, nausea or vomiting during ingestion of cleansing fluid.Though diet restriction with low-fiber diet is always advised to every screen before colonoscopy, the extent of diet restriction is widely variable and thus influences the degree of colon cleansing.

With commercialized low-residue diet (CLRD), diet restriction will be well controlled and variability of colon cleansing can be minimized such that guarantee a colonoscopy with good quality. In this RCT, we will compare the compliance of screen during colon cleansing using different protocol: namely 2000 ml PEG-ELS vs. 1500 ml plus low-residue diet.

DETAILED DESCRIPTION:
Setting: A multi-center study including the following teaching hospitals:

National Taiwan University Hospital, Taipei Taipei Medical University Hospital, Taipei E-Da Hospital, Kaohsiung Buddhist Tzu-Chi General Hospital, Taipei En Chu Kong Hospital, Taipei Far Eastern Memorial Hospital, Taipei

Study design: RCT, single blinded

Study subjects:

Inclusion criteria: Subjects who receives colonoscopy for screening or for clinical purpose Exclusion criteria: Subjects with polyposis, ileus, active GI bleeding, IBD, severe constipation, renal insufficiency, obesity with BMI≥30

Grouping: subjects will be randomized to the following groups:

1. Group A: 2000 ml PEG-ELS
2. Group B: 1500ml PEG-ELS with CLRD Randomization process: Random block sheet

Measurements:

1. Subjects who obey protocol or violate/withdraw protocol will be all recorded.
2. Parameters concerning patient compliance
3. Number of detected adenoma and their topographical distribution
4. Time required for A. Cecal intubation B. Overall procedure time
5. Colon cleansing effect evaluation

The degree of cleansing will be recorded individually for each bowel segment (rectum, sigmoid colon, descending colon, transverse colon, and ascending colon). Each segment will be rated using a 5-point scale: 4, very good-colon empty and clean; 3, good-presence of clear liquid in the gut; 2, moderate-presence of brown liquid or small amounts of semisolid residual stool, fully removable by suction or displaceable, thus allowing a complete visualization of the underlying mucosa; 1, bad-presence of semisolid stool, only partially removable with a risk of incomplete underlying mucosal visualization; and 0, very bad-presence of semisolid or solid stool, colonoscopy incomplete or has to be stopped. The overall quality of colonic cleansing will be based on the assessment of the individual segments using a scale of A, all segments clean (i.e., scores of 3 or 4 in all segments); B, residual brown liquid or suctionable semisolid stool (i.e., a score of 2) in at least one segment; C, partially removable stool preventing complete visualization of mucosa (i.e., a score of 1) in at least one segment; or D, at least one segment can not be examined due to the presence of solid stool (i.e., a score of 0). A grade of either A or B was defined, a priori, as successful colon cleansing.

Sample size estimation:

Assuming 80% power and significance level at 0.05, totally at least 112 cases will be required for each group (assuming 90% cases in 2000 ml achieving good or excellent preparation and 76% of 1500mL plus low-residue diet achieving the same cleansing effect).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who receives colonoscopy for screening or for clinical purpose

Exclusion Criteria:

* Subjects with polyposis, ileus, active GI bleeding, IBD, severe constipation, renal insufficiency, obesity with BMI≥30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Colon cleansing level | At the timing of colonoscopy

SECONDARY OUTCOMES:
adenoma detection rate | At the timing of colonoscopy
Cecal intubation time | At the timing of colonoscopy
Patient compliance including abdominal symptoms during colon cleansing, bowel movement on the way to hospital | -2hr
Whole procedural time | At the timing of colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Han-Mo Chiu, MD, Principal Investigator — National Taiwan University Hospital
Locations (5):
- Taiwan (5):
  - E-DA Hospital, Kaohsiung City
  - Buddhist Tzu-Chi General Hospital, Taipei
  - En Chu Kong Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei